CLINICAL TRIAL: NCT01008150
Title: A Phase II Randomized Clinical Trial Evaluating Neoadjuvant Therapy Regimens With Weekly Paclitaxel Plus Neratinib or Trastuzumab or Neratinib and Trastuzumab Followed by Doxorubicin and Cyclophosphamide With Postoperative Trastuzumab in Women With Locally Advanced HER2-Positive Breast Cancer
Brief Title: Phase II Randomized Trial Evaluating Neoadjuvant Therapy With Neratinib and/or Trastuzumab Followed by Postoperative Trastuzumab in Women With Locally Advanced HER2-positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-7
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant; neratinib; paclitaxel; trastuzumab; doxorubicin; cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; neratinib; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: paclitaxel + trastuzumab then A C (Active Comparator): 4 cycles of paclitaxel 80 mg/m2 on Days 1, 8, and 15 of a 28-day cycle. Trastuzumab concurrently with paclitaxel weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Following paclitaxel/trastuzumab, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm 2: paclitaxel + neratinib then A C (Experimental): 4 cycles of paclitaxel 80 mg/m2 on Days 1, 8, and 15 of a 28-day cycle. Neratinib 240 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Interventions: Drug: Paclitaxel; Drug: Neratinib; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm 3: paclitaxel + trastuzumab + neratinib then A C (Experimental): 4 cycles of paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle. Trastuzumab concurrently with paclitaxel, weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/trastuzumab/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Neratinib; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm 3 NR: paclitaxel+trastuzumab+neratinib (Experimental): Non-randomized: 4 cycles of paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle. Trastuzumab concurrently with paclitaxel, weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/trastuzumab/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Neratinib; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Arm 1: paclitaxel + trastuzumab then A C; Arm 3 NR: paclitaxel+trastuzumab+neratinib; Arm 3: paclitaxel + trastuzumab + neratinib then A C
Drug: Neratinib
  Arms: Arm 2: paclitaxel + neratinib then A C; Arm 3 NR: paclitaxel+trastuzumab+neratinib; Arm 3: paclitaxel + trastuzumab + neratinib then A C
Drug: Doxorubicin
  Other Names: Adriamycin; A
Drug: Cyclophosphamide
  Other Names: C

SUMMARY:
FB-7 is a Phase II, multi-center randomized study of neratinib in combination with weekly paclitaxel with or without trastuzumab followed by doxorubicin and cyclophosphamide (AC) as neoadjuvant therapy for women with HER2-positive locally advanced breast cancer. Patients in the control arm will receive neoadjuvant trastuzumab in combination with weekly paclitaxel followed by AC. The primary aim of the study is to determine the pathologic complete response (pCR) rate in breast and axillary nodes following the neoadjuvant therapy regimens. The secondary aims include determination of the pCR rate in breast only, clinical complete response (cCR) rate, two-year recurrence-free interval, two-year overall survival, toxicity of the neoadjuvant regimens, and exploration of molecular and genetic correlates of response.

DETAILED DESCRIPTION:
Sequential AC followed by a taxane initiated concurrently with trastuzumab has become a standard of care in the United States for operable HER2-positive breast cancer following initial surgery.

Trastuzumab, a recombinant humanized monoclonal antibody against the extracellular domain of the HER2 protein, was developed to block HER2 signaling pathways and has been shown to substantially improve the efficacy of chemotherapy in women with metastatic and early-stage HER2-positive breast cancers.

However, some patients develop recurrence and succumb to the disease following trastuzumab-based adjuvant therapy. Evaluation of additional approaches that target this pathway have shown promising results in trastuzumab-resistant breast cancer.

Neratinib (HKI-272), an orally administered small molecule, is an irreversible inhibitor of pan ErbB receptor tyrosine kinases, which distinguishes this small molecule from lapatinib. Because of the high degree of homology between kinase domains of EGFR and HER2, neratinib inhibits both EGFR and HER2 function. Neratinib is designed to block kinase activity by binding to the ATP site of the enzymes. In BT474 cell lines, HKI-272 effectively repressed phosphorylation of MAPK and Akt signal transduction pathways, whereas trastuzumab failed to completely inhibit HER2 receptor phosphorylation or downstream signaling events. In tumor xenografts which overexpress HER2, neratinib has been observed to repress tumor growth in a dose-dependent manner.

A comparison of overall response rates with lapatinib and neratinib in comparable patients, albeit in separate Phase II studies, suggest favorable efficacy of neratinib as monotherapy in trastuzumab-refractory patients (response rate of 5.1% vs. 26%) and in trastuzumab-naïve patients (response rate of 24% vs. 56%). Taken together, the data support the rationale that a small molecule TKI may be more efficacious than trastuzumab in the neoadjuvant setting, and that neratinib may be more active than lapatinib.

The study started as a two-arm design with randomization to the control arm (Arm 1) and to the investigational arm (Arm 2) in a 1:2 ratio. With the addition of a second investigation arm, (Arm 3), the study becomes a three-arm design with a 1:1:1 allocation ratio (about equal numbers of patients randomized to Arms 1, 2, and 3). The sample size will be up to 126 patients with about 42 evaluable patients in each arm. Patients who enter the trial but are not treated for any reason will be replaced. Accrual is expected to occur over 18 months. Patients will be randomized to one of three neoadjuvant therapy regimens: Patients in Arm 1 will receive 4 cycles of paclitaxel 80 mg/m2 administered on Days 1, 8, and 15 of a 28-day cycle. Trastuzumab will begin concurrently with paclitaxel and will be given weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Following paclitaxel/trastuzumab, standard AC will be administered every 21 days for 4 cycles; Patients in Arm 2 will receive 4 cycles of paclitaxel 80 mg/m2 administered on Days 1, 8, and 15 of a 28-day cycle. Neratinib 240 mg will be taken orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Standard AC administered every 21 days for 4 cycles will be administered following paclitaxel/neratinib therapy; Patients in Arm 3 will receive 4 cycles of paclitaxel 80 mg/m2 administered Days 1, 8, and 15 of a 28 day cycle with trastuzumab, beginning concurrently with paclitaxel, given weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg will be taken orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Standard AC will be administered every 21 days for 4 cycles following paclitaxel/trastuzumab/neratinib therapy.

In all arms, clinical response will be assessed by palpation between the chemotherapy regimens and prior to surgery. Following recovery from surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) will be administered every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy). Patients will receive adjuvant radiation therapy and endocrine therapy as clinically indicated.

At the time of local IRB approval of amendment #6, submission of fresh tumor samples for FB-7 correlative science studies will be optional for all patients. For patients who agree, a core biopsy procedure to procure three fresh tumor samples will be performed before randomization (after the patient has signed the consent form and has been screened for eligibility). Submission of a tumor block from the diagnostic core biopsy sample and a tumor block from gross residual disease greater than or equal to 1.0 cm, if found in the surgical specimen, will be required. In addition, a blood sample collected after randomization (before the start of study therapy) will also be required for the correlative science studies.

Beginning with Amendment #8, Arm 1 and Arm 2 were closed to accrual in the US subsequent to FDA approval of pertuzumab when given in combination with trastuzumab for neoadjuvant therapy in breast cancer. Pertuzumab and trastuzumab are both targeted therapy drugs. US patients enrolled in the study will not be randomized but will be placed into the combined targeted therapy group, Arm 3 NR, only. Randomization and study therapy for patients entered via institutions outside of the US remains unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a life expectancy of at least 10 years, excluding their diagnosis of breast cancer.
* Submission of a block from the diagnostic biopsy sample and from the surgical sample, if gross residual disease greater than or equal to 1.0 cm was removed at the time of surgery, is required for all patients
* Patients of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy and for at least 6 months after the last dose of study therapy.
* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1.
* Patients must have the ability to swallow oral medication.
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or by limited incisional biopsy.
* Patients must have ER analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then progesterone receptor (PgR) analysis must also be performed. (Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.)
* Breast cancer must be determined to be HER2-positive prior to randomization. Assays using FISH or CISH require gene amplification. Assays using IHC require a strongly positive (3+) staining score.
* Clinical staging, based on the assessment by physical exam, must be American Joint Committee on Cancer (AJCC) stage IIB, IIIA, IIIB, or IIIC: cT2 and cN1; cT3 and cN0 or cN1; Any cT and cN2 or cN3; or cT4
* The patient must have a mass in the breast or axilla measuring greater than or equal to 2.0 cm by physical exam, unless the patient has inflammatory breast cancer, in which case measurable disease by physical exam is not required.
* At the time of randomization, blood counts performed within 4 weeks prior to randomization must meet the following criteria: absolute neutrophil count (ANC) must be greater than or equal to 1200/mm3; Platelet count must be greater than or equal to 100,000/mm3; Hemoglobin must be greater than or equal to 10 g/dL
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to randomization must be met: total bilirubin must be less than or equal to upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and aspartate aminotransferase (AST) and ALT must be less than or equal to 1.5 x ULN for the lab.
* Patients with alkaline phosphatase greater than ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET, or PET-CT scan) performed within 4 weeks prior to randomization does not demonstrate metastatic disease and the requirements for adequate hepatic function are met.
* Patients with either unexplained skeletal pain or alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 4 weeks prior to randomization does not demonstrate metastatic disease. Patients with suspicious findings on bone scan or PET scan are eligible if suspicious findings are determined to be benign by x-ray, MRI, or biopsy.
* Serum creatinine performed within 4 weeks prior to randomization must be less than or equal to 1.5 x ULN for the lab.
* The left ventricular ejection fraction (LVEF) assessment by 2-D echocardiogram or multiple gated acquisition(MUGA) scan performed within 90 days prior to randomization must be greater than or equal to 50% regardless of the facility's LLN.

Exclusion Criteria:

* fine-needle aspiration (FNA) alone to diagnose the primary breast cancer.
* Excisional biopsy or lumpectomy performed prior to randomization.
* Surgical axillary staging procedure prior to randomization. (Procedures that are permitted prior to study entry include: 1) FNA or core biopsy of an axillary node for any patient, and 2) although not recommended, a pre-neoadjuvant therapy SN biopsy for patients with clinically negative axillary nodes.)
* Definitive clinical or radiologic evidence of metastatic disease. (Note: Chest imaging [mandatory for all patients] and other imaging [if required] must have been performed within 90 days prior to randomization.)
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral ductal carcinoma in situ (DCIS) treated with radiation therapy (RT). (Patients with a history of LCIS are eligible.)
* Contralateral invasive breast cancer at any time. (Patients with contralateral DCIS or lobular carcinoma in situ (LCIS) are eligible.)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to randomization.
* Known metastatic disease from any malignancy (solid tumor or hematologic).
* Previous therapy with anthracyclines, taxanes, cyclophosphamide, trastuzumab, or neratinib for any malignancy.
* Treatment including RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to randomization.
* Continued endocrine therapy such as raloxifene or tamoxifen (or other SERM) or an aromatase inhibitor. (Patients are eligible if these medications are discontinued prior to randomization.)
* Any continued sex hormonal therapy, e.g., birth control pills and ovarian hormone replacement therapy. Patients are eligible if these medications are discontinued prior to randomization.
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Intrinsic lung disease resulting in dyspnea.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Persistent greater than or equal to grade 2 diarrhea regardless of etiology.
* Sensory or motor neuropathy greater than or equal to grade 2, as defined by the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0.
* Conditions that would prohibit intermittent administration of corticosteroids for paclitaxel premedication.
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* Uncontrolled hypertension defined as a systolic BP greater than 150 mmHg or diastolic BP greater than 90 mmHg, with or without anti-hypertensive medications. (Patients with hypertension that is well-controlled on medication are eligible.)
* Cardiac disease (history of and/or active disease) that would preclude the use of any of the drugs included in the treatment regimen. This includes but is not confined to: Active cardiac disease: symptomatic angina pectoris within the past 180 days that required the initiation of or increase in anti-anginal medication or other intervention; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis. History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function; history of documented congestive heart failure (CHF); and documented cardiomyopathy.
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Pregnancy or lactation at the time of randomization.
* The investigator should assess the patient to determine if she has any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.
* Use of any investigational agent within 4 weeks prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-10; Primary Completion 2015-09 (Actual); Study Completion 2016-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (42):
- United States (30):
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente-San Diego, San Diego, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Edward Cancer Center, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - Yorkville Family Practice, Yorkville, Illinois
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Missouri-Ellis Fischel, Columbia, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University Hospital and Medical Center - SUNY Stony Brook, Stony Brook, New York
  - CCOP Carolinas HealthCare System, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western Reserve University/University Hospitals of Cleveland, Cleveland, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roper Hosp & Med Asso (Care Alliance Health), Charleston, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - West Virginia University Hospitals Inc., Morgantown, West Virginia
- Canada (3):
  - University of Montreal Hospital Group, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Azienda Ospedaliera Fatebenefratelli Milano, Milan, Italy
- MBCCOP - San Juan, San Juan, Puerto Rico
- Spain (7):
  - Galicia Hospital Universitario A Coruña, A Coruña, Galicia
  - Madrid Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Cataluna Hospital del Mar, Barcelona
  - Cataluna Hospital Quiron de Barcelona, Barcelona
  - Extremadura Hospital San Pedro Alcantara, Cáceres
  - Cataluna Hospital Amau de Vilanova de Lleida, Lleida
  - Valencia Institut Valencia de Oncologia, Valencia

REFERENCES:
- [Derived] Jacobs SA, Robidoux A, Abraham J, Perez-Garcia JM, La Verde N, Orcutt JM, Cazzaniga ME, Piette F, Antolin S, Aguirre E, Cortes J, Llombart-Cussac A, Di Cosimo S, Kim RS, Feng H, Lipchik C, Lucas PC, Srinivasan A, Wang Y, Song N, Gavin PG, Balousek AD, Paik S, Allegra CJ, Wolmark N, Pogue-Geile KL. NSABP FB-7: a phase II randomized neoadjuvant trial with paclitaxel + trastuzumab and/or neratinib followed by chemotherapy and postoperative trastuzumab in HER2+ breast cancer. Breast Cancer Res. 2019 Dec 3;21(1):133. doi: 10.1186/s13058-019-1196-y. PMID 31796073
- [Derived] Jankowitz RC, Abraham J, Tan AR, Limentani SA, Tierno MB, Adamson LM, Buyse M, Wolmark N, Jacobs SA. Safety and efficacy of neratinib in combination with weekly paclitaxel and trastuzumab in women with metastatic HER2-positive breast cancer: an NSABP Foundation Research Program phase I study. Cancer Chemother Pharmacol. 2013 Dec;72(6):1205-12. doi: 10.1007/s00280-013-2262-2. PMID 24077916

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Paclitaxel + Trastuzumab Then A C: 4 cycles of paclitaxel 80 mg/m2 on Days 1, 8, and 15 of a 28-day cycle. Trastuzumab concurrently with paclitaxel weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Following paclitaxel/trastuzumab, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Paclitaxel
  Trastuzumab
  Doxorubicin
  Cyclophosphamide
- Arm 2: Paclitaxel + Neratinib Then A C: 4 cycles of paclitaxel 80 mg/m2 on Days 1, 8, and 15 of a 28-day cycle. Neratinib 240 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Paclitaxel
  Neratinib
  Doxorubicin
  Cyclophosphamide
- Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C; Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then AC: 4 cycles of paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle. Trastuzumab concurrently with paclitaxel, weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/trastuzumab/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Paclitaxel
  Trastuzumab
  Neratinib
  Doxorubicin
  Cyclophosphamide
Period: Overall Study
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then AC
Started | 43 | 43 | 43 | 12
Completed | 42 | 42 | 42 | 12
Not Completed | 1 | 1 | 1 | 0
Not completed — did not receive study drug | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C: 4 cycles of paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle. Trastuzumab concurrently with paclitaxel, weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/trastuzumab/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Paclitaxel
  Trastuzumab
  Neratinib
  Doxorubicin
  Cyclophosphamide
- Total: Total of all reporting groups
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C | Total
Number analyzed (Participants) | 42 | 42 | 42 | 12 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.70) | 53.7 (9.87) | 50.9 (12.68) | 48.7 (11.94) | 51.6 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 42 | 12 | 138
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 4 | 1 | 15
  Not Hispanic or Latino | 38 | 35 | 38 | 8 | 119
  Unknown or Not Reported | 1 | 0 | 0 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 34 | 38 | 7 | 116
  Black or African American | 3 | 4 | 3 | 2 | 12
  Asian | 2 | 3 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White/American Indian or Alaskan Native | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response in Breast and Axillary Lymph Nodes.
Description: Number of participants with no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes after neoadjuvant chemotherapy
Time Frame: At time of surgery, approximately 7 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm 3 NR: Paclitaxel + Trastuzumab + Neratininb Then AC: 4 cycles of paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle. Trastuzumab concurrently with paclitaxel, weekly for a total of 16 doses (4 mg/kg loading dose, then 2 mg/kg weekly). Neratinib 200 mg orally once daily beginning on Day 1 of paclitaxel and continuing through Day 28 of the final cycle of paclitaxel. Following paclitaxel/trastuzumab/neratinib therapy, standard AC every 21 days for 4 cycles. Following surgery, trastuzumab (8 mg/kg loading dose, then 6 mg/kg) every 3 weeks to complete 1 year of targeted therapy (either preoperative trastuzumab therapy or neratinib therapy)
  Paclitaxel
  Trastuzumab
  Neratinib
  Doxorubicin
  Cyclophosphamide
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratininb Then AC
Number analyzed (Participants) | 42 | 42 | 42 | 12
Participants | 16 | 14 | 21 | 5

2. Secondary Outcome: Pathologic Complete Response in Breast.
Description: Number of participants with by no histologic evidence of invasive tumor cells in the surgical breast specimen.
Time Frame: At time of surgery, approximately 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C
Number analyzed (Participants) | 42 | 42 | 42 | 12
Participants | 21 | 16 | 22 | 6

3. Secondary Outcome: Clinical Complete Response, as Measured by Physical Exam
Description: Upon physical exam the number of participants with resolution of all target and non-target lesions identified at baseline and no new lesions or other signs of disease progression.
Time Frame: At the completion of AC prior to surgery, approximately 7 months
Population: Only patients with palpable disease at baseline are included in this outcome. Arm1-38 patients at baseline, 2 patients missing data. Arm 2-35 patients at baseline, 4 patients missing data. Arm 3-38 patients at baseline, 4 patients missing data. Arm 3 NR-10 patients at baseline, 1 patient missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C
Number analyzed (Participants) | 36 | 31 | 34 | 9
Participants | 25 | 25 | 28 | 6

4. Secondary Outcome: Recurrence-free Interval (RFI)
Description: Number of participants with no events of inoperable progressive disease and local, regional and distant recurrence.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C
Number analyzed (Participants) | 42 | 42 | 42 | 12
Participants | 42 | 39 | 40 | 12

5. Secondary Outcome: Overall Survival
Description: Number of participants alive at 24 months.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C
Number analyzed (Participants) | 42 | 42 | 42 | 12
Participants | 42 | 42 | 42 | 12

6. Secondary Outcome: Adverse Events Experienced by Participants as a Measure of Toxicity
Description: Number of patients with at least one adverse event.
Time Frame: Assessed through 2 years from randomization
Population: Refer to Adverse Events section for more details.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then A C
Number analyzed (Participants) | 42 | 42 | 42 | 12
Participants | 41 | 42 | 42 | 12

ADVERSE EVENTS:
Arm/Group | Arm 1: Paclitaxel + Trastuzumab Then A C | Arm 2: Paclitaxel + Neratinib Then A C | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then AC
Serious Adverse Events (participants affected / at risk) | 7/42 | 7/42 | 10/42 | 2/12
Other Adverse Events (participants affected / at risk) | 41/42 | 42/42 | 42/42 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Paclitaxel + Trastuzumab Then A C (N=42) | Arm 2: Paclitaxel + Neratinib Then A C (N=42) | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C (N=42) | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then AC (N=12)
Infection (Infections and infestations) | 1 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 2 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Left venrticular dysfunction (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Paclitaxel + Trastuzumab Then A C (N=42) | Arm 2: Paclitaxel + Neratinib Then A C (N=42) | Arm 3: Paclitaxel + Trastuzumab + Neratinib Then A C (N=42) | Arm 3 NR: Paclitaxel + Trastuzumab + Neratinib Then AC (N=12)
Diarrhoea (Gastrointestinal disorders) | 16 | 42 | 41 | 12
Nausea (Gastrointestinal disorders) | 12 | 25 | 20 | 8
Vomiting (Gastrointestinal disorders) | 7 | 16 | 13 | 6
Constipation (Gastrointestinal disorders) | 6 | 12 | 11 | 7
Dyspepsia (Gastrointestinal disorders) | 9 | 13 | 6 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 6 | 7 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Oral pain (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 18 | 22 | 18 | 8
Asthenia (General disorders) | 9 | 7 | 10 | 0
Pain (General disorders) | 4 | 9 | 5 | 2
Pyrexia (General disorders) | 1 | 6 | 6 | 3
Oedema peripheral (General disorders) | 2 | 5 | 3 | 2
Catheter site pain (General disorders) | 1 | 1 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 3 | 1
Chills (General disorders) | 0 | 2 | 1 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 7 | 3 | 8 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 22 | 15 | 6
Rash (Skin and subcutaneous tissue disorders) | 9 | 9 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 3
Dermatitis aceniform (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 7 | 16 | 17 | 7
Aspartate aminotransferase increased (Investigations) | 6 | 13 | 14 | 7
Neutraphil count (Investigations) | 5 | 6 | 1 | 0
Weight decreased (Investigations) | 2 | 6 | 4 | 3
White blood cell count (Investigations) | 5 | 4 | 1 | 1
Haemoglobin (Investigations) | 2 | 5 | 2 | 2
Alanine aminotransferase (Investigations) | 2 | 2 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 4 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0 | 0
Blood alkaline phosphatase (Investigations) | 1 | 2 | 0 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 10 | 7 | 7 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 8 | 4 | 3
Dysgeusia (Nervous system disorders) | 3 | 8 | 7 | 3
Dizziness (Nervous system disorders) | 4 | 5 | 6 | 4
Neurapathy peripheral (Nervous system disorders) | 6 | 5 | 3 | 0
Paraesthesia (Nervous system disorders) | 4 | 4 | 5 | 1
Neurotoxicity (Nervous system disorders) | 2 | 1 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 4 | 1
Restless leg syndrome (Nervous system disorders) | 2 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 2 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 13 | 9 | 8 | 3
Anaemia (Blood and lymphatic system disorders) | 9 | 5 | 8 | 2
Leukopenia (Blood and lymphatic system disorders) | 5 | 6 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 11 | 11 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 8 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 7 | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 5 | 4 | 0
Dehyrdration (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 5 | 2 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2 | 1
Influenza (Infections and infestations) | 2 | 0 | 3 | 0
Folliculitis (Infections and infestations) | 3 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 6 | 3 | 3
Anxiety (Psychiatric disorders) | 4 | 5 | 4 | 0
Mood altered (Psychiatric disorders) | 2 | 4 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 3 | 6 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 3 | 3 | 0
Dry eye (Eye disorders) | 0 | 2 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 7 | 8 | 2 | 0
Embolism (Vascular disorders) | 0 | 4 | 1 | 1
Flushing (Vascular disorders) | 1 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 3 | 3 | 2 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 5 | 6 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 4 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less